CLINICAL TRIAL: NCT06032507
Title: Effect of High-pressure Pulsatile Lavage Versus Manual Rinsing on Bone Cement Penetration in Total Knee Arthroplasty - A Randomized Clinical Trial
Brief Title: Effect of High-pressure Pulsatile Lavage Versus Manual Rinsing on Bone Cement Penetration in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIBSP-HPL-2021-90
Record Dates: First submitted 2022-02-23; First posted 2023-09-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2023-09

CONDITIONS: Knee
Keywords: Total Knee Arthroplasty Cementation; Bone cement penetration; High Pressure Pulsatile Lavage; Pulsatile lavage; Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: 100 patients undergoing primary TKA
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed lavagegroup (Experimental): Bone cementation with previous high-pressure pulsatile lavage
  Interventions: Procedure: Bone lavage previous to cementation
- Non-pulsed lavage group (Experimental): Bone cementation with previous manual rinsing lavage
  Interventions: Procedure: Bone lavage previous to cementation

INTERVENTIONS:
Procedure: Bone lavage previous to cementation — Bone lavage previous to cementation in total knee arthroplasty

SUMMARY:
Background

Bone irrigation is essential in cemented total knee arthroplasty surgical technique in order to improve cement penetration and interdigitation into cancellous bone, that is going to determine the strength of the bone-cement interface.

Purpose

To report the effect of high-pressure pulsatile lavage versus manual rinsing on bone cement penetration in total knee arthroplasty.

Methods

This is a single-centre, prospective, randomized, controlled clinical trial. The study included 100 patients undergoing primary total knee arthroplasty. All patients meeting inclusion criteria were randomly assigned to the pulsed lavage or non-pulsed lavage group. The cumulative bone cement penetration was radiologically assessed in antero posterior and lateral radiograph views in 10 zones according to the Knee Society Scoring System. A statistical analysis was performed between both groups comparing bone cement penetration cumulative scores.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years
* Age <89 years
* Clinical symptoms of knee osteoarthritis
* Failed conservative treatment

Exclusion Criteria:

* Metal allergies
* Active or latent knee sepsis
* Extensor mechanism dysfunction
* Morbid obesity
* Several peripheral vascular disease
* Noncompliance due to major psychiatric or neurological disorders.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Cumulative bone cement penetration | 48 hours postoperative xrays
  The cumulative bone cement penetration was radiologically assessed in AP and lateral radiograph views in 10 zones according to the Knee Society Scoring System (for each zone, <4 = nonprogressive, 5-9 = risk of progression, >10 = risk of failure) - minimum 0, maximum non established-.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharkey PF, Hozack WJ, Rothman RH, Shastri S, Jacoby SM. Insall Award paper. Why are total knee arthroplasties failing today? Clin Orthop Relat Res. 2002 Nov;(404):7-13. doi: 10.1097/00003086-200211000-00003. PMID 12439231
- [Background] Peters CL, Craig MA, Mohr RA, Bachus KN. Tibial component fixation with cement: full- versus surface-cementation techniques. Clin Orthop Relat Res. 2003 Apr;(409):158-68. doi: 10.1097/01.blo.0000058638.94987.20. PMID 12671498
- [Background] Maistrelli GL, Antonelli L, Fornasier V, Mahomed N. Cement penetration with pulsed lavage versus syringe irrigation in total knee arthroplasty. Clin Orthop Relat Res. 1995 Mar;(312):261-5. PMID 7634612
- [Background] Clarius M, Seeger JB, Jaeger S, Mohr G, Bitsch RG. The importance of pulsed lavage on interface temperature and ligament tension force in cemented unicompartmental knee arthroplasty. Clin Biomech (Bristol). 2012 May;27(4):372-6. doi: 10.1016/j.clinbiomech.2011.10.006. Epub 2011 Nov 1. PMID 22051198
- [Background] Jaeger S, Seeger JB, Schuld C, Bitsch RG, Clarius M. Tibial cementing in UKA: a three-dimensional analysis of the bone cement implant interface and the effect of bone lavage. J Arthroplasty. 2013 Oct;28(9 Suppl):191-4. doi: 10.1016/j.arth.2013.05.014. Epub 2013 Jun 21. PMID 23790498
- [Background] Ritter MA, Herbst SA, Keating EM, Faris PM. Radiolucency at the bone-cement interface in total knee replacement. The effects of bone-surface preparation and cement technique. J Bone Joint Surg Am. 1994 Jan;76(1):60-5. doi: 10.2106/00004623-199401000-00008. PMID 8288666
- [Background] Ewald FC. The Knee Society total knee arthroplasty roentgenographic evaluation and scoring system. Clin Orthop Relat Res. 1989 Nov;(248):9-12. PMID 2805502
- [Background] Wing N, Van Zyl N, Wing M, Corrigan R, Loch A, Wall C. Reliability of three radiographic classification systems for knee osteoarthritis among observers of different experience levels. Skeletal Radiol. 2021 Feb;50(2):399-405. doi: 10.1007/s00256-020-03551-4. Epub 2020 Aug 11. PMID 32780155
- [Background] Schlegel UJ, Bishop NE, Puschel K, Morlock MM, Nagel K. Comparison of different cement application techniques for tibial component fixation in TKA. Int Orthop. 2015 Jan;39(1):47-54. doi: 10.1007/s00264-014-2468-x. Epub 2014 Aug 1. PMID 25082179
- [Derived] Ramirez-Bermejo E, Fa-Binefa M, Pilco-Inga J, Jordan-Sales M, Aguilera-Roig X, Gonzalez-Rodriguez JC. Effect of high-pressure pulsatile lavage versus manual rinsing on bone cement penetration in total knee arthroplasty: a randomized clinical trial. Knee Surg Relat Res. 2025 Nov 4;37(1):47. doi: 10.1186/s43019-025-00298-x. PMID 41188974